CLINICAL TRIAL: NCT01537315
Title: Hydroxychloroquine in Cardiovascular Disease in Patients With Chronic Kidney Disease: A Proof of Concept Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 132036
Record Dates: First submitted 2012-02-10; First posted 2012-02-23 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Kidney Failure, Chronic; Cardiovascular Disease; Arteriosclerosis
Keywords: Kidney Failure, Chronic; Cardiovascular Disease; Arteriosclerosis
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases; Arteriosclerosis | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Matching Placebo (Placebo Comparator): Patients with cardiovascular disease (CVD) and chronic kidney disease (CKD) will be randomized to either hydroxychloroquine (HCQ) or matching placebo in a 3:1 ratio (approximately 39 to HCQ and 13 to placebo)
  Interventions: Other: Matching Placebo
- Hydroxychloroquine (Experimental): Patients with cardiovascular disease (CVD) and chronic kidney disease (CKD) will be randomized to either hydroxychloroquine (HCQ) or matching placebo in a 3:1 ratio (approximately 39 to HCQ and 13 to placebo)
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — 200 mg capsule daily for 10 +/- 4 days, then 200 mg twice daily till end of study (duration approximately 6 months)
  Other Names: Plaquenil
  Arms: Hydroxychloroquine
Other: Matching Placebo — matching placebo capsule 200 mg daily for 10 +/- 4 days and thereafter 200 mg twice a day for duration of study, approximately 6 months
  Arms: Matching Placebo

SUMMARY:
Presence of multiple traditional and nontraditional risk factors of atherosclerosis and cardiovascular disease (CVD) including inflammation in patients with chronic kidney disease (CKD) contribute to high CVD morbidity and mortality in this patient population. Additionally, the traditional approaches towards the therapy of CVD have little impact on CV mortality in these patients. Hydroxychloroquine (HCQ) used as anti-inflammatory in rheumatological disorders, has multiple beneficial properties relevant to the process of vascular disease. The effects of HCQ on atherosclerosis (AS) and vascular disease in CKD is not known yet. Thus, the study hypothesis is that HCQ treatment in individuals with CKD will provide clinically significant benefit in the management of CVD and will provide biological and functional atherosclerotic benefits.

DETAILED DESCRIPTION:
This pilot study has been designed to look at the impact of hydroxychloroquine (HCQ) in the clinical model of accelerated atherosclerosis (AS) in the chronic kidney disease (CKD) population. This intervention is designed to have an impact on the initiation and progression of AS by reducing systemic inflammation, improving or restoring vascular endothelial function, and by improving the milieu of metabolic syndrome and insulin resistance.

The current study is a proof of concept study for the expansion of the use of HCQ for a new indication for the treatment of AS and cardiovascular disease (CVD) in patients with CKD.University of Arkansas for Medical Sciences (UAMS) has filed an Investigational New Drug (IND) for a new indication on 4/28/11. The FDA responded that this study is exempt from an IND.

This "Proof-of-Concept" randomized double blinded placebo controlled study will evaluate the nature and extent of HCQ effects, and if found significantly beneficial, it will be used to guide the development of a large, multicenter, randomized control trial of HCQ to examine the hard clinical end points of CVD and mortality in patients with advanced CKD. The investigators propose to enroll 62 subjects to achieve the effects of HCQ in 52 individuals (39 HCQ group and 13 placebo group).

ELIGIBILITY:
Inclusion Criteria:

* Measured stage IV proteinuric chronic kidney disease with an estimated Modification of Diet in Renal Disease (MDRD) GFR (eGFR) of 18 to 35 ml/min.
* Current or history of documented proteinuria of more than or equal to 300 mg/dL in 24 hours or a spot urine protein to creatinine ratio of greater than 0.3 ug/mg.
* Not on dialysis.
* Ages 18 to 80 years, both sexes, all races and ethnicities

Exclusion Criteria:

* glucose-6-phosphate dehydrogenase (G6PD) deficiency or known hypersensitivity to 4-aminoquinoline compounds (such as chloroquine or hydroxychloroquine).
* Abnormal liver functions; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) more than 2.5 times the normal or international normalized ratio (INR) without being anti-coagulated greater than 1.4.
* Known chronic active infections like HIV, Hepatitis B or Hepatitis C positive, chronic osteomyelitis etc.
* Recent serious infection including Pneumonia requiring hospitalization, meningitis, septicemia in the 2 months prior to screening.
* Active or recently treated (< 1 year in remission) malignancy or systemic inflammatory diseases (Patients with localized squamous cell carcinoma of the skin are eligible).
* Pregnancy, breastfeeding or planning to become pregnant during the course of the study.
* Use of systemic corticosteroids or other immunosuppression within last 3 months (acute course of steroid for a gouty arthritis or chronic obstructive pulmonary disease (COPD) is eligible if > 1 month ago).
* History of prolonged corrected QT interval > 450.
* Inability to attend or comply with treatment or follow-up scheduling.
* Life expectancy less than 6 months or uncontrolled congestive heart failure (CHF) (defined as more than 2 admissions in prior 6 months).
* Any other condition the PI determines may put the research subject in jeopardy during the course of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dumitru Rotaru, MD, Principal Investigator — University of Arkansas
Locations (3):
- United States (3):
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Florida, Gainesville, Florida

RESULTS

PARTICIPANT FLOW:
Groups:
- Matching Placebo: Patients with CVD and CKD will be randomized to either hydroxychloroquine (HCQ) or placebo in a 3:1 ratio (approximately 39 to HCQ and 13 to placebo)
  Placebo comparator: matching capsule 200 mg daily for 10 +/- 4 days and thereafter 200 mg twice a day for duration of study, approximately 6 months
- Hydroxychloroquine: Patients with CVD and CKD will be randomized to either hydroxychloroquine (HCQ) or placebo in a 3:1 ratio (approximately 39 to HCQ and 13 to placebo)
  Hydroxychloroquine: 200 mg capsule daily for 10 +/- 4 days, then 200 mg twice daily till end of study (duration approximately 6 months)
Period: Overall Study
Arm/Group | Matching Placebo | Hydroxychloroquine
Started | 1 | 7
Completed | 1 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Matching Placebo | Hydroxychloroquine | Total
Number analyzed (Participants) | 1 | 7 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 6 | 7
Region of Enrollment [Number; unit: participants]
  United States | 1 | 7 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Inflammatory Marker, Hs-C Reactive Protein, at 6 Months
Description: Hs-CRP will be measured at baseline (before study drug) and at end of study (6 months). This marker is measured by ELISA assay from serum.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Matching Placebo: Patients with cardiovascular disease (CVD) and chronic kidney disease (CKD) will be randomized to either hydroxychloroquine (HCQ) or placebo in a 3:1 ratio (approximately 39 to HCQ and 13 to placebo)
  Placebo comparator: matching placebo capsule 200 mg daily for 10 +/- 4 days and thereafter 200 mg twice a day for duration of study, approximately 6 months
Arm/Group | Matching Placebo | Hydroxychloroquine
Number analyzed (Participants) | 1 | 7
ng/ml | 18653.6 (NA) — Standard deviation not calculated because only one participant was assessed. | 14825.8 (12416.8)
Statistical Analysis 1: Comparison: Hydroxychloroquine; Test type: Superiority or Other; p = 0.4521, ANOVA — A paired comparison between baseline CRP values with values obtained after 1, 3, and 6 months of treatment was conducted, with a p-value of 0.05 used as the a priori threshold of statistical significance

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Matching Placebo | Hydroxychloroquine
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/7
Other Adverse Events (participants affected / at risk) | 0/1 | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matching Placebo (N=1) | Hydroxychloroquine (N=7)
Stomach upset (Gastrointestinal disorders) | 0 (0) | 2 (2) — 2 subjects reported upset stomach which resolved for both.
Increased Blood Pressure (Cardiac disorders) | 0 (0) | 1 (1) — Increased blood pressure in one subject which was treated with higher dose of antihypertensive

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No